CLINICAL TRIAL: NCT00915265
Title: Continuous Preperitoneal Versus Epidural Infusion of Local Anesthetic for Enhanced Postoperative Recovery Following Open Colorectal Surgery
Brief Title: Continuous Preperitoneal Infusion of Local Anesthetic (CPA) Versus Epidural Infusion of Local Anesthetic (EA) in Fast-Track Open Colorectal Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0052
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Open Colorectal Surgery; Early Rehabilitation After Surgery
Keywords: Epidural analgesia; Continuous preperitoneal analgesia; Surgery; Open colorectal surgery; Fast-track surgery; ERAS

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Other: Multilobed catheter (group CPA) — - CPA group: continuous preperitoneal administration of 0.2% ropivacaine using a multilobed catheter positioned between the previously closed parietal peritoneum and the underside of the transversalis fascia
Other: Multilobed catheter (group EA) — EA group : thoracic epidural infusion of 0.2 % ropivacaine

SUMMARY:
The purpose of this study is to compare the continuous preperitoneal infusion of local anesthetic and continuous epidural analgesia for postoperative pain management in fast-track open colorectal surgery.

DETAILED DESCRIPTION:
Optimized pain relief allowing early mobilization is a prerequisite for enhanced recovery after surgery. Open colorectal surgery is associated with severe and prolonged postoperative pain, especially during mobilization. No analgesic technique has fulfilled all requirements of optimal efficacy: no side effects, low costs, high patient compliance, and improvement in outcome, and consequently, multimodal analgesic techniques have been introduced with a focus on opioid sparing to improve analgesia and recovery. Epidural analgesia (EA) has shown a marked benefit in controlling pain at mobilization, and significantly improves pain management when compared with systemic patient-controlled morphine analgesia. However, eligible patients may not benefit from it because of technical problems or failure of efficiency. Recently, continuous preperitoneal infusion of local anesthetic (CPA) has been shown to be an effective method to relief pain after open colorectal surgery, to reduced morphine consumption and accelerated postoperative recovery. However, this technique has never been evaluated in a fast-track program (ERAS protocol). Moreover, continuous preperitoneal infusions of local anesthetic and epidural analgesia have never been compared.

The purpose of this randomized and double-blinded study is to compare these two techniques on pain control during mobilization, as a prerequisite for enhanced recovery after open colorectal surgery: 1- CPA group: continuous preperitoneal administration of 0.2% ropivacaine using a multilobed catheter positioned between the previously closed parietal peritoneum and the underside of the transversalis fascia + intravenous morphine (patient-controlled analgesia, PCA) as a rescue; 2- EA group: epidural infusion of 0.2% ropivacaine (patient-controlled epidural analgesia, PCEA) + continuous preperitoneal administration of 0.9% saline.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Open colorectal surgery through a midline incision with a primary anastomosis
* American Society of Anesthesiologists (ASA) physical status I to III

Exclusion Criteria:

* Obesity (body mass index > 35 kg/m2)
* Pregnancy
* Inflammatory bowel diseases
* Contraindication for epidural analgesia (patient refusal, active sepsis, coagulopathy)
* Chronic renal failure (with creatinin clearance < 30 ml/min)
* Significant hepatic failure (prothrombin ratio < 50%, factor V < 50%)
* Chronic pain
* Preoperative opioid consumption
* Preoperative cognitive dysfunction
* Preoperative psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-10; Primary Completion 2018-07 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Pain measured at mobilization (defined as pain experienced during transition from supine to the sitting position) using the visual analogue pain scale (VAS) from 0 (no pain) to 10 (worst pain imaginable), at 24 hour after tracheal extubation (H0) | at 24 hour after tracheal extubation (H0)

SECONDARY OUTCOMES:
Duration of Post-Anesthesia Care Unit (PACU) stay | in the post-anesthesia care unit

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel FUTIER, MD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Jouve P, Bazin JE, Petit A, Minville V, Gerard A, Buc E, Dupre A, Kwiatkowski F, Constantin JM, Futier E. Epidural versus continuous preperitoneal analgesia during fast-track open colorectal surgery: a randomized controlled trial. Anesthesiology. 2013 Mar;118(3):622-30. doi: 10.1097/ALN.0b013e3182800d94. PMID 23426208